CLINICAL TRIAL: NCT00620308
Title: A Human Physiologic Study to Evaluate the Renal and Neurohumoral Effects of a Novel Chimeric Natriuretic Peptide, CD-NP, in Subjects With Stable Chronic Heart Failure
Brief Title: CD-NP in Subjects With Stable Chronic Heart Failure
Acronym: CD-NP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John A. Schirger, John Schirger ,MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 07-005523
Record Dates: First submitted 2008-02-10; First posted 2008-02-21 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-08

CONDITIONS: Stable Chronic Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CD-NP low-dose study drug (Experimental)
  Interventions: Drug: CD-NP
- CD-NP high-dose study drug (Experimental)
  Interventions: Drug: CD-NP
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CD-NP — One of two dosage levels (20 ng/kg/min and another level to be finalized) as a continuous intravenous infusion for four hours
  Arms: CD-NP high-dose study drug; CD-NP low-dose study drug
Drug: Placebo — Dextrose 5% in water (the vehicle)
  Arms: Placebo

SUMMARY:
This human physiologic study will evaluate the effects of a new drug called CD-NP in individuals with stable chronic heart failure, with a focus on evaluating responses of the kidneys and the hormonal system.

DETAILED DESCRIPTION:
CD-NP is a novel chimeric natriuretic peptide which was created by combining the 22 amino acids of human C-type natriuretic peptide (CNP) and the 15-amino-acid C-terminus of Dendroaspis natriuretic peptide (DNP). The rationale for selecting CNP, a natriuretic peptide of endothelial cell origin, is that it exhibits predominantly venodilating effects, which may minimize systemic hypotension. Moreover, its anti-proliferative action is also a highly desirable property for novel cardiovascular drugs. However, a limitation of CNP is that it does not exert significant renal actions, whereas, DNP is potently natriuretic and diuretic. Thus, CD-NP was synthesized with the goal of combining the above complementary profiles of CNP and DNP into a single chimeric peptide.

ELIGIBILITY:
Inclusion Criteria:

1. Male and non-pregnant female subjects, aged 21 or above, with stable chronic HF of primary cardiac etiology, resting left ventricular ejection fraction (LVEF) ≤ 40 % documented within the last 2 years, and New York Heart Association functional class I - III symptoms
2. Be willing to provide informed consent.

Exclusion Criteria:

1. Known allergy or other adverse reactions to exogenous natriuretic peptides (CD-NP or its components, nesiritide, other natriuretic peptides, or related compounds).
2. Women who are pregnant, or breast-feeding.
3. Having received nesiritide for within 7 days prior to prior to entry into the study.
4. Having received any investigational drug or device within 30 days prior to entry into the study.
5. Clinically unstable patients (e.g. systolic blood pressure < 90 mmHg, ongoing requirement for vasopressors or mechanical circulatory support, or mechanical ventilation).
6. Recent hospitalization for decompensated HF or recent defibrillation for cardiac resuscitation within 30 days prior to randomization.
7. Prior organ transplantation, being on a waiting list for organ transplantation, or ongoing requirement for longterm vasoactive support.
8. Patients with guarded prognosis who are unlikely to derive meaningful benefit from CD-NP.
9. Use of sulfonamides, non-steroidal anti-inflammatory drugs, probenecid, or other drugs that are known to alter renal function within 5 half-lives prior to the first dose of CD-NP or placebo.
10. Presence of cardiac lesions or comorbidities that may contraindicate the use of natriuretic peptides, such as clinically significant cardiac valvular stenosis, hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, primary pulmonary hypertension, or uncorrected congenital heart disease that contraindicates the use of vasodilators.
11. History of blood pressure > 190/115 mmHg or unexplained syncope within the past 3 months.
12. Symptomatic carotid artery disease, known critical carotid stenosis, or stroke within the past 3 months
13. Clinically significant renal artery stenosis
14. Baseline hemoglobin < 10.0 g/dL.
15. Serum sodium < 130 mEq/L, potassium < 3.6 mEq/L, or magnesium < 1.7 mEq/L.
16. Elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) at least 5 times the upper limit of normal or bilirubin at least 3 times the upper limit of normal
17. Creatinine clearance (CrCl) < 50 ml.min-1.1.73m-2, as calculated by Cockcroft-Gault formula and adjusted for body surface area within the past year or at screening, or requirement for dialysis.
18. History of alcohol abuse within the past 6 months.
19. Consumption of a phosphodiesterase-5 inhibitor (sildenafil, vardenafil, or tadalafil) within 72 hours of receiving CD-NP or placebo.
20. Inability to communicate effectively with study personnel.
21. bmi>38

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
To assess renal, neurohumoral and non-invasive hemodynamic physiologic parameters | Within the first 24 to 36 hours of the study and at follow-up visits (days 9 and 30)

CONTACTS AND LOCATIONS:
Overall Officials: John C. Burnett, Jr., MD, Study Director — Mayo Foundation
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States